CLINICAL TRIAL: NCT06555835
Title: Effect of Lower Extremity Flexibility on Postural Stability
Brief Title: Effect of Flexibility on Postural Stability
Status: Recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Atlas University (Other)
Responsible Party: Principal Investigator, Kübra Alpay, Lecturer of Pysiotherapy and Rehabilitation Department, Bezmialem Vakif University
Other Study IDs: Ka24-3
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postural stability has an important role for functional movements, injury prevention and the performance of many athletic skills. Therefore, it is very important to understand the factors that affect postural stability. The aim of this study is to investigate the effect of lower extremity flexibility on postural stability in healthy individuals.

DETAILED DESCRIPTION:
Postural stability provides the relationship between the body's center of gravity and the base of support using somatosensory information. Postural stability is a very important determinant for functional movements. It is known that postural stability plays an important role in the performance of many sports skills, protection from injuries and daily life activities. Therefore, it is very important to understand the factors affecting postural stability well.

Joint range of motion, muscle strength and flexibility are among the factors affecting postural stability. Hip, knee and ankle joint movements controlled along the kinetic chain are important in providing postural stability. The aim of the study is to evaluate the effect of lower extremity flexibility on dynamic postural stability in healthy individuals. Healthy volunteers between the ages of 18-25 will be included in the study and flexibility and postural stability assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-25
* Volunteering to participate in the study

Exclusion Criteria:

* Having a diagnosis of neurological, orthopedic, vestibular, rheumatological disorder
* Having a history of musculoskeletal injury or surgery within the last year
* Participating in a regular exercise program

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population will consist of healthy young adults who meet inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-10-25 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Passive straight leg raise test | Baseline
  Test is performed in the supine position. Measurement of hip flexion angle is performed with a universal goniometer at the end point of the movement.
Passive ankle dorsiflexion range of motion | Baseline
  During the measurement, individuals are in a supine position. The ankle joint range of motion measurement is performed with a universal goniometer.
Postural stability | Baseline
  Biodex Balance System (Biodex Medical Systems, Inc. USA) will be used in the dynamic single leg stance test and sensory integration of balance clinical test evaluations. Lower scores indicate better stability and higher scores mean poor balance.

CONTACTS AND LOCATIONS:
Overall Officials: Kubra Alpay, PhD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)